CLINICAL TRIAL: NCT04111822
Title: Pilot Study on the Use of Hydrocortisone, Vitamin c and Tiamine in Patient With Sepsis and Septic Shock
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cristina Martinez (Other)
Responsible Party: Sponsor-Investigator, Cristina Martinez, Master in Science and clinical reseracher manager, Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta
Organization: Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT number 2018-000196-32
Record Dates: First submitted 2019-08-05; First posted 2019-10-01 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Sepsis; Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional treatment of septic shock (Active Comparator): Conventional treatment of septic shock according to current management guidelines
  Interventions: Drug: on crystalloid fluid and Tranexamic acid
- Current management plus ascorbic acyd,thiamine and vitamin C (Experimental): Conventional treatment of septic shock according to current management guidelines associated with:
  i. Hydrocortisone 50 mg every 6 hours for 7 days or until discharge from the ICU with subsequent withdrawal in descending pattern for 3 days ii. Vitamin C (ascorbic acid) 1.5 gr diluted in 100 ml of 5% SG every 6 hours for 4 days (16 doses) iii. Thiamine 200 mg diluted in 100 ml of SG 5% or SF 0.9% every 12 hours for 4 days iv. Measurement of vitamin C levels prior to administration of the first dose of vitamin C
  Interventions: Drug: red blood cells transfusion, tranexamic acid (TXA) and fibrinogen concentrate

INTERVENTIONS:
Drug: red blood cells transfusion, tranexamic acid (TXA) and fibrinogen concentrate — Phase III, randomized, multicenter, open-label and parallel group pilot study, which aims to study mortality at 28 days of admission in patients with septic shock treated with usual management and patients treated with ascorbic acid, thiamine and hydrocortisone added to usual driving
  Other Names: experimental intervention
  Arms: Current management plus ascorbic acyd,thiamine and vitamin C
Drug: on crystalloid fluid and Tranexamic acid — Resuscitation with crystalloids, Performing culture battery, antibiotic therapy
  Other Names: clinical practice intervention
  Arms: Conventional treatment of septic shock

SUMMARY:
Due to the high incidence, mortality and short and long term complications of sepsis and septic shock, it is necessary to look for strategies to try to minimize this impact.

DETAILED DESCRIPTION:
Based on the current literature, we can affirm that the decrease in ascorbic acid levels in patients with sepsis and septic shock is directly proportional to the evolution to multiorgan failure and inversely proportional to survival. After assessing the safety in the administration of ascorbic acid as well as the decrease or almost abolition of its impact at the renal level after the association of thiamine, and the synergy provided by the administration of hydrocortisone, it is decided to implement the "Metabolic Resucitation Protocol" and assess its impact on our septic patients

ELIGIBILITY:
Inclusion Criteria:

* Patients> 18 years of age with diagnosis of septic shock and multiorgan failure admitted to our Unit
* Entry into the ICU once diagnosed with sepsis and / or septic shock. The first 24 hours after admission to the ICU will be established as an inclusion limit
* Written informed consent.

Exclusion Criteria:

* Patients under 18
* Pregnancy
* Coexistence of other types of shock at admission
* Limitation of therapeutic effort or ICT (Conditional Intensive Therapy) upon admission to the ICU. It refers to patients in whom, prior to admission to the ICU, it was decided not to perform any or some of the usual treatment measures for sepsis, or in which a time limit is established in which in case of non-response they would withdraw intensive measures. This limitation will be indicated by your treating physician and if it exists, the patient would be excluded from the study.
* Patient with a history of previous intake of ascorbic acid, thiamine or corticosteroids in the month prior to admission to the ICU
* Patients considered immunodeficient (More than 10 mg of prednisone or its equivalent per day in the last 2 weeks, immunosuppressive therapy or diagnosis of acquired immunodeficiency syndrome).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Estimate and compare hospital survival after 28 days of admission in patients with septic shock treated with usual management and patients treated with ascorbic acid, thiamine and hydrocortisone added to usual management | 28 days
  Number of patients that are alive after 28 days of admission
Compare mortality at 7, 14 and 28 days after admission in patients with septic shock treated with usual management and patients treated with ascorbic acid, thiamine and hydrocortisone added to usual management. | 28 days
  Number of patients that are exitus at 7, 14 and 28 days after admission

SECONDARY OUTCOMES:
Compare the days of admission to the ICU in patients with septic shock treated with usual management and patients treated with ascorbic acid, thiamine and hydrocortisone added to usual management. | 28 days
  number of days that patient stay in ICU department
Compare the days of mechanical ventilation in patients with septic shock treated with usual management and patients treated with ascorbic acid, thiamine and hydrocortisone added to usual management | 28 days
  compare the days of use of mechanical ventilation in every arm
Compare the days of need for vasoactive drug requirements and doses in patients with septic shock treated with usual management and patients treated with ascorbic acid, thiamine and hydrocortisone added to usual management. | 28 days
  compare the days of need for vasoactive drug requirements in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Juliana Gonzalez, MD, Principal Investigator — Hospital Dr Josep Trueta
Locations (1):
- Hospital Dr Josep Trueta, Girona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gonzalez Londono J, Vera Ching C, Sebastian Cernuda P, Morales Pedrosa JM, Lorencio C, Sirvent JM. Effect of vitamin C, thiamine and hydrocortisone in critically ill septic patients. The Metabolic Resus RCT. Med Intensiva (Engl Ed). 2024 Apr;48(4):238-240. doi: 10.1016/j.medine.2023.11.002. Epub 2023 Nov 18. No abstract available. PMID 37985341